CLINICAL TRIAL: NCT01277549
Title: Evaluation of the Spectra Optia® Apheresis System Mononuclear Cell (MNC) Collection Procedure in Healthy Blood Donors
Status: Completed | Type: Observational
Sponsor: Terumo BCT (Industry)
Collaborators: Versiti Blood Health (Other); Key Biologics, LLC (Industry); LeukoLab (Unknown); Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: BCT10-03
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Leukapheresis
Keywords: Leukapheresis; Hematopoetic Stem Cell Mobilization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-mobilized donors: In this arm the collection efficiency of mononuclear cells from non-mobilized donors will be studied.
  Interventions: Device: Mononuclear cell collection.
- G-CSF mobilized donors: In this arm the collection efficiency of CD34+ cells will be studied.
  Interventions: Device: Mononuclear cell collection.

INTERVENTIONS:
Device: Mononuclear cell collection. — Each donor will undergo one apheresis procedure to collect mononuclear cells from their peripheral blood.

SUMMARY:
The purpose of this protocol is to characterize the performance of CaridianBCT's Spectra Optia Apheresis System, when used to collect mononuclear cells (MNCs) and cluster of differentiation 34 (CD34) positive cells from healthy nonmobilized blood donors and healthy G-CSF (granulocyte colony stimulating factor) mobilized blood donors, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Acceptable health history to allow blood product collection
* Weight >50<125 Kg (kilogram).
* Male or non-pregnant, non-nursing female.
* General good health, as determined by questionnaire.
* Normal prescreening complete blood count.
* Platelet count>150 x 10^3/uL (microliter) at initial screening and >120 x 10^3/uL immediately prior to leukapheresis.
* Adequate peripheral venous access to allow collection of product.
* Able to read, understand, and sign the informed consent form. Additional Inclusion Criteria for Mobilized Subjects
* If male, be willing to use a condom during sexual relations with a female partner until 48 hours following the last G-CSF injection.
* If female and of childbearing potential, be willing to use a medically acceptable contraceptive until 48 hours following the last G-CSF injection.

Exclusion Criteria:

* a) Collection or loss of:

  * more than a ½ pint (1 cup) of whole blood within the prior 56 days or,
  * more than 3 L (liter) of whole blood or 1.5 L of red blood cells within the prior 12 months or,
  * more than 12 L of plasma within the prior 12 months or,
  * a leukapheresis within the prior six weeks or,
  * a plateletpheresis within the prior 48 hours or two within the prior 7 days or twenty-four within the last 12 months or,
  * a plasmapheresis within the prior 48 hours or two within the prior 7 days.
* Acute or symptomatic chronic lung disease.
* Active or chronic heart disease, including hypertension controlled by medication.
* History of hematologic malignancy or chronic hematologic disorder or bleeding disorder.
* Reactive test indicative of infection with T. pallidum, Human T-lymphotropic virus, HIV, Hepatitis C Virus, or Hepatitis B Virus (except isolated Hepatitis B Core Antibody Reactivity.
* Presence of psychological traits or physiological or medical conditions that would make subject unlikely to tolerate the procedures.
* Subjects taking prescription medications other than those deemed allowable by the investigator.
* Abnormal serum electrolytes or serum calcium levels.
* Abnormal serum creatinine level.
* Abnormal liver function results on ALT (alanine amino transferase) test.
* Abnormal coagulation testing on prothrombin time or partial thromboplastin time.
* Inadequate antecubital veins for leukapheresis or inability or unwillingness to tolerate leukapheresis.
* If female, pregnant or lactating. Additional Exclusion Criteria for Mobilized Subjects
* Received a G-CSF injection in the prior 4 months, or received more than twenty-five (25) doses of G-CSF (a dose includes several individual injections administered on one occasion).
* Known hypersensitivity to G-CSF or any E. coli-derived products.
* History of autoimmune condition or disorder, unless approved by principal investigator.
* Immediate family history (parents, grandparents, siblings, children) of hematologic malignancy.
* Active or history of iritis (anterior uveitis) or episcleritis.
* History of deep vein thrombosis or pulmonary embolism.
* Current treatment with lithium.
* Spleen tip palpable during physical exam.
* Positive SickleDex test.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Community Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome R Bill, MD, Study Director — Terumo BCT
Locations (3):
- United States (3):
  - Leukolab/Allcells, Emeryville, California
  - Key Biologics, Memphis, Tennessee
  - Blood Center of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult donors were recruited at three blood collection centers to undergo a mononuclear cell collection using the experimental device, between January and September, 2011.
Groups:
- G-CSF Mobilized Donors: In this arm the donors received G-CSF (granulocyte colony stimulating factor) prior to the MNC (mononuclear cell) collection. G-CSF causes the mobilization of hematopoetic stem cells which are CD34 (cluster of differentiation 34) + to the peripheral blood. Collection efficiency of all mononuclear cells and of the CD34+ subset of mononuclear cells was assessed.
- Non-mobilized Donors: In this arm, donors were not mobilized prior to mononuclear cell collection. Only collection efficiency of mononuclear cells could be assessed as CD34+ cells are not present in this population.
Period: Overall Study
Arm/Group | G-CSF Mobilized Donors | Non-mobilized Donors
Started | 41 | 29
Completed | 15 | 15
Not Completed | 26 | 14
Not completed — Failed to meet eligibility criteria | 13 | 9
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 10 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: Data is given only for subjects who completed the study. Reasons why subjects did not complete the study are given above in Participant Flow.
Groups:
- G-CSF Mobilized Donors: Donors received G-CSF prior to MNC collection
- Nonmobilized Donors: Donors not mobilized prior to MNC collection
- Total: Total of all reporting groups
Arm/Group | G-CSF Mobilized Donors | Nonmobilized Donors | Total
Number analyzed (Participants) | 15 | 15 | 30
Age Continuous [Median (Full Range); unit: Years of Age] — Median and range reported are for donors who completed the study.
  Years of Age | 25 [19 to 45] | 33 [29 to 47] | 31 [19 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mononuclear Cell Collection Efficiency
Description: The collection efficiency for a given cell type is defined as the percent of processed cells of that cell type that are in fact collected.
Time Frame: One day
Population: Results are given for all per protocol subjects.
Measure: Median (Full Range); unit: % of processed MNCs that were collected
Groups:
- Nonmobilized Donors: Donors were not mobilized prior to MNC collection.
Arm/Group | G-CSF Mobilized Donors | Nonmobilized Donors
Number analyzed (Participants) | 15 | 15
% of processed MNCs that were collected | 61 [17 to 147] | 57 [27 to 92]

2. Secondary Outcome: Platelet Collection Efficiency
Description: Platelet contamination of the cell product was measured as the platelet collection efficiency, that is, as the percent of platelets processed that were collected.
Time Frame: One Day
Population: Per protocol
Measure: Median (Full Range); unit: % of processed platelets collected
Groups:
- G-CSF Mobilized Donors: In this arm, donors were mobilized with G-CSF prior to collection.
- Nonmobilized Donors: In this arm, donors were not mobilized prior to collection.
Arm/Group | G-CSF Mobilized Donors | Nonmobilized Donors
Number analyzed (Participants) | 15 | 15
% of processed platelets collected | 19 [12 to 47] | 12 [5 to 21]

3. Secondary Outcome: Hematocrit of MNC Product
Description: The hematocrit of the collected product was used to quantitate RBC (red blood cell) contamination.
Time Frame: One Day
Population: Per protocol
Measure: Median (Full Range); unit: RBC % of product volume
Arm/Group | G-CSF Mobilized Donors | Nonmobilized Donors
Number analyzed (Participants) | 15 | 15
RBC % of product volume | 4.0 [1.4 to 6.0] | 4.0 [2.0 to 5.0]

4. Secondary Outcome: Granulocyte % of MNC Product
Description: Granulocyte contamination of the MNC product was quantitated as the percent of total product WBC (white blood cell) that were segmented granulocytes or bands.
Time Frame: One day
Population: Results given for all per protocol subjects.
Measure: Median (Full Range); unit: percentage of WBCs collected
Arm/Group | G-CSF Mobilized Donors | Nonmobilized Donors
Number analyzed (Participants) | 15 | 15
percentage of WBCs collected | 15.0 [0.0 to 48] | 1.7 [0.3 to 9.0]

5. Secondary Outcome: Viability of the Collected MNC Product
Description: The viability of the collected white blood cells was assessed using the 7-AAD (7-amino actinomycin D) viability dye in a flow cytometric assay. Viability assessment is incorporated into the CD34 assay. This assay was only performed on G-CSF mobilized donors as nonmobilized donor have too few CD34+ cells to detect. Thus viability of the collected WBCs is reported only for the G-CSF mobilized arm.
Time Frame: One day
Population: Per Protocol
Measure: Median (Full Range); unit: percentage of total WBCs collected
Arm/Group | G-CSF Mobilized Donors
Number analyzed (Participants) | 15
percentage of total WBCs collected | 99 [90 to 100]

6. Primary Outcome: CD34+ Cell Collection Efficiency
Description: The collection efficiency for CD34+ cells is defined as the percent of processed CD34+ cells that were in fact collected.
Time Frame: one day
Population: Results are given for all per protocol subjects.
Measure: Median (Full Range); unit: % of processed CD34+ cells collected
Arm/Group | G-CSF Mobilized Donors
Number analyzed (Participants) | 15
% of processed CD34+ cells collected | 77 [43 to 111]

ADVERSE EVENTS:
Time Frame: For the Nonmobilized Arm, adverse events were collected during the leukapheresis procedure itself and for one week following the procedure. For the G-CSF mobilized arm, adverse events were also collected during the 5 days of mobilization.
Description: All subjects who underwent a leukapheresis procedure were included in the adverse event analysis. This includes the categories "COMPLETED" and "NOT COMPLETED--Protocol Violation" on the Participant Flow section above. Thus 15+10=25 Mobilized and 15+1+16 Nonmobilized subjects are included for a total of 41 subjects.
Groups:
- Nonmobilized Donors: Donors not mobilized prior to MNC collection. Note that some Adverse Events (Flu-like symptoms, Muscle Aches, and Bone Pain) apply only to G-CSF mobilized donors. Nonmobilized donors were not assessed for these adverse events as they were not "at risk".
Arm/Group | G-CSF Mobilized Donors | Nonmobilized Donors
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/16
Other Adverse Events (participants affected / at risk) | 19/25 | 8/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | G-CSF Mobilized Donors (N=25) | Nonmobilized Donors (N=16)
Arm numbness/stiffness (General disorders) | 0 (0) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0/0 (0)
Citrate reaction (General disorders) | 6 (6) | 5 (5)
Flu-like symptoms (General disorders) | 10 (10) | 0/0 (0)
Muscle Aches (General disorders) | 12 (12) | 0/0 (0)
Nausea (General disorders) | 0 (0) | 2 (2)
Venous infiltration/hematoma (General disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less